CLINICAL TRIAL: NCT04954807
Title: Growth and Body Composition of Low Birth Weight Infants Supplemented With Human Milk Fortifier After Discharge: A Double-Blind Randomized Clinical Trial
Brief Title: Indonesia After Discharge LBW Infant HMF Supplementation Study
Acronym: DAHLIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, yoga devaera, Head of Division of Nutrition and Metabolic Diseases of Child Health Dept, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-02-0127
Record Dates: First submitted 2021-06-14; First posted 2021-07-08 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Low; Birthweight; Breast Feeding, Exclusive; Gestational Age and Weight Conditions
Keywords: Low Birth Weight; Breast Feeding; Body Mass Index; Human Milk Fortifier; Small Gestational Age
MeSH Terms: conditions — Birth Weight; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Subjects in the intervention group will be given the new human milk fortifier which contains protein, lipid, carbohydrate and micronutrients while the control group will receive placebo (polysaccharides 0.9 g/1 g placebo and maltose 0.1 g/1 g placebo and minerals). Assuming the average weight is 2 Kg, 6 scoops (@1.0 g) will provide 1.95 g protein and 25.5 Kcal in the intervention group while 6 scoops of 1.1 g in the control group will provide 26.4 Kcal with no protein. Three times a day, supplementation with 2.0 gram (intervention group) or 2.2 gram (control group) of study product will be provided, regardless of the actual weight of the subject.
  Both groups will receive iron supplementation 2 drops daily (5 mg elemental iron in forms of Fe III hydroxide polymaltose complex) since 2 month old as a routine supplementation recommended by Indonesian Pediatrics Society.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One investigator who do not involve in recruitment and outcome measures will generate randomization list by computer application and set up the list into Redcap randomization set up. No one except him will know the sequence of randomization. Research assistant will randomize subjects into one of four group according to Redcap assignment. The manufacturer prepare the study product into four groups: A,B,C,D and kept the code until the statistical analysis completed. All investigators, care providers and study subjects aware of the active or placebo group. Research assistants who recruit the study subject are not allowed to open the tin. One research assistant who does no meet study subject will measure the weight of tin before and after the supplementation.
  Subject only meet with researchers individually and will not meet other subjects so they will not know the content of the other tin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Milk Fortifier (Active Comparator): human milk fortifier which contains protein, lipid, carbohydrate and micronutrients
  Interventions: Dietary Supplement: human milk fortified
- placebo (Placebo Comparator): Placebo is made of polysaccharides (0.9 g/1 g placebo) and maltose (0.1 g/1 g placebo) and minerals.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: human milk fortified — HMF will be given 6 scoops a day
  Arms: Human Milk Fortifier
Dietary Supplement: placebo — Placebo will be given six scoops a day
  Arms: placebo

SUMMARY:
Low birth weight (LBW) infant (1800-2449 gram) will be given the new human milk fortifier (HMF) which contains protein, lipid, carbohydrate and micronutrients after discharge. Human Milk Fortifier or placebo (carbohydrate only with similar calorie content) will be provided until 3 months of age. The investigators want to evaluate if the addition of HMF to mother's milk while breastfeeding LBW infants after discharge influences growth and body composition up to 3 months of age.

DETAILED DESCRIPTION:
This is a prospective two arms parallel double-blind randomized clinical trial in LBW infants. Clinically healthy LBW infants discharge on oral feeding of human milk before 2 weeks of age (< 15 days old) will be invited to participate in the study. Exclusively or predominantly breastfed infants will be encourage to use finger feeding as method of supplementation, but mothers can choose their own preferences if they wish to do so.

After signing the informed consent by parent, subject will be randomized to one of four group. Randomization list were prepare by one investigator who do not involve in recruitment, outcome measures and statistical analysis. Study product will be labeled as A, B, C D in similar tin. Only manufacturer know the content of these tins and the code will be revealed after statistical analysis completed. Parents will be given this 200 g tin of study product and ask to return the tin after 14 days of opening. Unblinded assistant will weight the tin before and after opening to estimate the HMF intake for 14 days.

This study will be conducted in several hospitals in Greater Jakarta.

Adherence to study protocol will be encouraged during face to face session initially in dispensing study product and subsequent visits (visit 1 at one-month-old, visit 2 at two months old). These sessions will include the reminder of the importance of following study protocol, breastfeeding support if needed and discussion about difficulties that arise. The investigators will also remind mothers via text to fill in three days diary of intake one week before each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Low birth weight infants (1800-2499 g) with oral feeding
2. Exclusively breastfed or predominantly breastfed (consuming term infant formula less than 50 ml/Kg BW/day) at discharge
3. Discharge from the hospital before 2 weeks of age and maximal age of enrolment is 14 days old
4. Live in greater Jakarta
5. Parents agree in writing to study participation and indicate their intention to follow study procedures.

Exclusion Criteria:

Any subject who has major congenital anomaly or any other disorder(s) that infers with normal feeding, growth, and neurodevelopment.

Participating in another intervention trial

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Gaining weight | three months of age
  Gain in weight (g/kg initial weight & difference) between study enrolment and three months of age

SECONDARY OUTCOMES:
Average weight gain | enrollment to three months of age
  Average daily weight gain (g/kg/day) from enrolment to at three months of age
Gaining length | Three months of age
  Gain in length (mm initial length & difference) from study enrolment to the age of 3 months
Head circumference | Three months of age
  Gain in head circumference (mm initial head circumference & difference) from study enrolment to the age of 3 months
Weight for age | Three months of age
  Difference of weight for age (Z score) from study enrolment to the age of 3 months
Body fat percentage | Three months of age
  Difference in body fat percentage between groups
Stool consistency | enrollment to three months of age
  Median type of stools according to Diapered Infant stool chart between groups
Stool frequency | enrollment to three months of age
  average stool frequency per day between groups
Vomit | enrollment to three months of age
  Number of subjects who reported to have vomit between groups
Bloating | enrollment to three months of age
  Number of subjects who reported to experience bloating between groups
Fever | enrollment to three months of age
  Number of subjects who reported to experience fever between groups
Rehospitalization | enrollment to three months of age
  Number of subjects who reported being hospitalized between groups

CONTACTS AND LOCATIONS:
Overall Officials: Yoga Devaera, MD, Principal Investigator — Indonesia University
Locations (4):
- Indonesia (4):
  - Budi Kemuliaan Hospital, Jakarta, Central Jakarta
  - Hermina Hospital, Bekasi, West Java
  - Pasarebo Regional Hospital, Jakarta
  - Koja District Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be published in a scientific journal. Others data will be available upon request to principle investigator.
Supporting Information: Study Protocol
Time Frame: Upon acceptance in scientific journal in one year from data completion
Access Criteria: Open access according to the journal